CLINICAL TRIAL: NCT03158558
Title: Multi-Couple Group Intervention for PTSD
Brief Title: Intensive Weekend Retreat Multi-Couple Group Therapy for PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); US Department of Veterans Affairs (U.S. Federal Agency); The University of Texas Health Science Center at San Antonio (Other); The Citadel (Unknown); Toronto Metropolitan University (Other); University of Denver (Other); Duke University (Other); VA Boston Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Steffany J Fredman, Ph.D., Assistant Professor of Human Development and Family Studies, Penn State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC20160094H
Record Dates: First submitted 2017-05-15; First posted 2017-05-18 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AM-CBCT for PTSD (Experimental): Accelerated, Multi-Couple Group Cognitive-Behavioral Conjoint Therapy delivered in a single weekend retreat
  Interventions: Behavioral: Accelerated, Multi-Couple Group CBCT for PTSD

INTERVENTIONS:
Behavioral: Accelerated, Multi-Couple Group CBCT for PTSD — Intensive weekend retreat version of cognitive-behavioral conjoint therapy for PTSD (Monson & Fredman, 2012)
  Other Names: AM-CBCT for PTSD

SUMMARY:
The purpose of this study is to test an intensive, multi-couple group version of a couple therapy for PTSD delivered to active duty Service Members or Veterans with PTSD and their romantic partners in a single weekend retreat. The study will be conducted on or near Fort Hood in Kileen, Texas. Twenty-four couples will be treated with this therapy and assessed immediately before treatment, 1 month after treatment, and 3 months after treatment.

DETAILED DESCRIPTION:
Numerous studies have documented an association between posttraumatic stress disorder (PTSD) symptoms and intimate relationship problems in both Service Members and Veterans and their partners, including relationship distress, physical and psychological aggression, and psychological distress in partners. In prior work, the investigators have demonstrated that cognitive-behavioral conjoint therapy for PTSD (CBCT for PTSD), a 15-session couple-based therapy for PTSD, is efficacious in simultaneously treating PTSD and comorbid symptoms and improving intimate relationship functioning. However, the current format of fifteen 75-minute sessions over 15 weeks presents challenges for large-scale dissemination for active duty Service Members and recently discharged Veterans who have deployed in support of 9/11.

The purpose of this uncontrolled trial is to pilot a brief, scalable version of CBCT for PTSD in which session content is taught in an accelerated, multi-couple group format (AM-CBCT for PTSD) that has the potential for rapid dissemination and implementation, while capturing the majority of the benefits of the original therapy format. Accelerated, multi-couple group CBCT for PTSD (AM-CBCT for PTSD) will be delivered in a single weekend retreat to 24 active duty Service Members and recently discharged Veterans with PTSD who have deployed post-9/11 and their partners. Participants will be assessed at pre-treatment, one month after treatment, and 3 months after treatment.

The study seeks to answer the following questions:

1. Will accelerated, multi-couple group CBCT for PTSD delivered in a weekend retreat (AM-CBCT for PTSD) be associated with significant improvements in clinician-rated PTSD symptom severity, as measured by the Clinician-Administered PTSD Scale for DSM-5 (CAPS-5), one month after treatment and at 3-month follow-up?
2. Will accelerated, multi-couple group CBCT for PTSD delivered in a weekend retreat (AM-CBCT for PTSD) be associated with significant improvements in secondary outcomes (e.g., patient self-reported PTSD and comorbid symptom severity, relationship satisfaction), one month after treatment and at 3-month follow-up?

ELIGIBILITY:
Inclusion Criteria:

* Married or cohabitating couples who have been together the past 3 months in which one partner is a Service Member or recently discharged Veterans eligible for treatment at Carl R. Darnall Army Medical Center (CRDAMC) with PTSD who has deployed since 9/11, seeking treatment for PTSD.
* Diagnosis of PTSD as determined by the Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) and a CAPS-5 score > 25. The Service Member or Veteran with PTSD must have experienced a Criterion A event that is a specific combat-related event or high magnitude operational experience that occurred during a military deployment in support of combat operations following 9/11. The diagnosis of PTSD may be indexed to that event or to another Criterion A event.
* Both individuals must be able to speak and read English.

Exclusion Criteria:

* Couple is separated and/or has taken steps to dissolve their relationship (e.g., divorce)
* Currently participating in evidence-based treatment for PTSD (Prolonged Exposure, Cognitive Processing Therapy, or Cognitive-Behavioral Conjoint Therapy for PTSD).
* Recent manic episode (past 12 months) or a psychotic disorder (as determined by the Mania and Psychosis modules of the MINI)
* Current alcohol dependence (as determined by an a score of ≥ 4 on items #4-6 and a total score of ≥20 on the AUDIT)
* Evidence of a moderate or severe traumatic brain injury (as determined by the inability to comprehend the baseline screening questionnaires)
* Current suicidal ideation severe enough to warrant immediate attention (as determined by the Depressive Symptoms Index - Suicidality Subscale; DSI-SS)
* Evidence or admission of severe intimate aggression as indicated by a "yes" endorsement to the one-question Screen for Conflict Question by either member of the couple occurring within the past 6-months.
* Partner who meets diagnostic criteria for PTSD according to the Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) or PTSD Checklist - Stressor Specific (PCL-S).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Clinician Administered PTSD Scale (CAPS-5) | change in PTSD symptoms at 1 and 3 months posttreatment
  semi-structured clinician interview to determine presence and severity of PTSD symptoms

SECONDARY OUTCOMES:
PTSD Checklist for DSM-5 (PCL-5) | change in PTSD symptoms at 1 and 3 months posttreatment
  patient self-report rating of PTSD symptom severity
Patient Health Questionnaire-9 (PHQ-9) | change in PTSD symptoms at 1 and 3 months posttreatment
  self-report measure of depressive symptom severity
Couples Satisfaction Index (CSI) | change in relationship satisfaction at 1 and 3 months posttreatment
  self-report measure of relationship satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Steffany J. Fredman, Ph.D., Principal Investigator — The Pennsylvania State University
Locations (1):
- University of Texas Health Sciences Center San Antonio, Killeen, Texas, United States

IPD SHARING:
Plan to Share IPD: No